CLINICAL TRIAL: NCT03552536
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti- Retroviral Activity of MK-8583 Monotherapy in Anti-Retroviral Therapy (ART)-Naïve, HIV-1 Infected Patients
Brief Title: MK-8583 Single Dose Study in Human Immunodeficiency Virus Type 1 (HIV-1) Infected Participants (MK-8583-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8583-002; 2017-004017-92 (EudraCT Number); MK-8583-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A: MK-8583 100mg (Experimental): After fasting, a single oral dose of 100 mg MK-8583 in capsule form.
  Interventions: Drug: MK-8583
- B: MK-8583 ≤ 150 mg (Experimental): After fasting, a single oral dose of ≤ 150 mg MK-8583 in capsule form, with the dose based on the results from earlier treatments
  Interventions: Drug: MK-8583
- C: MK-8583 ≤ 150 mg (Experimental): After fasting, a single oral dose of ≤ 150 mg MK-8583 in capsule form, with the dose based on the results from earlier treatments
  Interventions: Drug: MK-8583

INTERVENTIONS:
Drug: MK-8583 — A single oral dose of MK-8583 in capsule form

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics (PK), and anti-retroviral therapy (ART) activity of the tenofovir prodrug, MK-8583 monotherapy in ART-naïve, HIV-1 infected participants. The primary hypothesis is that at a dose that is sufficiently safe and generally well tolerated, MK-8583 has superior anti-retroviral activity compared to historical placebo, as measured by change from baseline in plasma HIV-1 ribonucleic acid (RNA) (log10 copies/mL) at 168 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male with female partner(s) of child-bearing potential use required methods of birth control.
* Female of reproductive potential must demonstrate a nongravid state at the pretrial (screening) visit and agree to use acceptable methods of birth control beginning at the pretrial (screening) visit, throughout the trial and until 30 days following cessation of treatment.
* Postmenopausal female, defined as without menses for at least 1 year and have a documented follicle stimulating hormone (FSH) level in the postmenopausal range at pretrial (screening).
* Surgically sterile female's status is post hysterectomy or oophorectomy.
* Is documented HIV-1 positive
* Is diagnosed with HIV-1 infection ≥ 3 months prior to screening.
* Is ART-naïve, defined as having never received any anti-retroviral agent; or ≤ 30 consecutive days of an investigational anti-retroviral agent, excluding a nucleoside reverse transcriptase inhibitor (NRTI), or ≤ 60 consecutive days of combination ART not including a NRTI.

Exclusion Criteria:

* Is mentally or legally institutionalized/incapacitated, has significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder over the last 5 years.
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a history of cancer (malignancy).
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Is positive for Hepatitis B surface antigen.
* Has a history of chronic Hepatitis C unless there has been documented cure.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
* Has participated in another investigational trial within 4 weeks or 5 half-lives, whichever is greater, prior to the pre-trial (screening) visit.
* Uses or anticipates using any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of trial drug, throughout the trial, until the post-trial visit.
* Consumes greater than 3 glasses of alcoholic beverages, wine or distilled spirits per day.
* Consumes excessive amounts of caffeinated beverages per day.
* Is an excessive smoker (i.e., more than 10 cigarettes/day) and is unwilling to restrict smoking to ≤10 cigarettes per day.
* Has a positive urine drug screen (except for cannabis) at screening and/or pre-dose.
* Has received any investigational agent or any anti-retroviral agent within 60 days of study drug administration; or intends to receive any ART during this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Charite Research Organisation GmbH ( Site 0001), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with human immunodeficiency virus-1 (HIV-1) infection who were naïve to anti-retroviral therapy (ART) were enrolled. Only participants from Panel A were recruited. Due to an earlier than anticipated achievement of the study objectives, a decision was made not to conduct Panels B and C.
Groups:
- B: MK-8583 ≤ 150 mg; C: MK-8583 ≤ 150 mg: After fasting, a single oral dose of ≤ 150 mg MK-8583 in capsule form.
Period: Overall Study
Arm/Group | A: MK-8583 100mg | B: MK-8583 ≤ 150 mg | C: MK-8583 ≤ 150 mg
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants from Panel A were recruited. Due to an earlier than anticipated achievement of the study objectives, a decision was made not to conduct Panels B and C.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: MK-8583 100mg | B: MK-8583 ≤ 150 mg | C: MK-8583 ≤ 150 mg | Total
Number analyzed (Participants) | 5 | 0 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (10.9) |  |  | 30.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 0 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 0 | 0 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Day 29
Population: All participants who received at least one dose of treatment. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
Participants | 4

2. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Change From Baseline in Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) at 168 Hours Post-dose.
Description: Plasma HIV-1 RNA was measured at baseline and 168 hours after dosing. Change from baseline for MK-8583 at 168 hours post-baseline was estimated from longitudinal data analysis (LDA) model containing fixed effects for time (predose, 168 hours postdose) and a random effect for participant. The change from baseline in plasma HIV-1 RNA in participants administered MK-8583 was compared with historical placebo data.
Time Frame: Baseline (pre-dose) and 168 hours post-dose.
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
log10 copies/mL | -0.63 [-1.30 to 0.05]
Statistical Analysis 1: Comparison: A: MK-8583 100mg; Test type: Superiority — Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a longitudinal data analysis (LDA) model containing fixed effects for study and time, and a random effect for participants. Least squares (LS) mean (95% confidence interval) for change from baseline at 168 hours post dose of pooled historical placebo was -0.03 log10 copies/mL (-0.14, 0.09); Posterior Mean Difference = -0.60 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8583 and placebo at least 0.5 log10 copies/mL was 64%

4. Secondary Outcome: Area Under the Concentration Time Curve From Time 0-168 Hours Postdose (AUC0-168hr) of Tenofovir Diphosphate (TFV-DP)
Description: Values of TFV-DP in peripheral blood mononuclear cells (PBMCs) were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The area under the concentration time curve from time 0-168 hours post-dose (AUC0-168hr) for intracellular TFV-DP is presented.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, and 168 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr*nmol/L | 324000 (179)

5. Secondary Outcome: Time to Achieve Maximum Concentration (Tmax) of TFV-DP
Description: Values of TFV-DP in PBMCs were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The time to achieve maximum concentration (Tmax) of intracellular TFV-DP is presented.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 312 and 672 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr. | 12 [4 to 12]

6. Secondary Outcome: Maximum Concentration (Cmax) of TFV-DP
Description: Values of TFV-DP in PBMCs were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The maximum concentration (Cmax) of intracellular TFV-DP is presented.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 312 and 672 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
nmol/L | 4660 (182)

7. Secondary Outcome: Concentration at 168 Hours Postdose (C168hr) of TFV-DP
Description: Values of TFV-DP in PBMCs were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The concentration at 168 hours postdose (C168hr) of TFV-DP is presented. It is hypothesized that the true geometric mean (GM) of TFV-DP in PBMC is ≥ 0.1 μM (100 nmol/L).
Time Frame: 168 hr postdose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment. The PBMC sample from one participant was processed incorrectly, so was not included in the analysis. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 4
nmol/L | 940 (414)

8. Secondary Outcome: Apparent Terminal Half-life (t1/2) of TFV-DP
Description: Values of TFV-DP in PBMCs were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The apparent terminal half-life (t1/2) of intracellular TFV-DP is presented.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 312 and 672 hours postdose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment. One participant who had insufficient data on terminal phase was not included in the analysis. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 4
hr. | 241 (23.7)

9. Secondary Outcome: Area Under the Concentration Time Curve From Time 0-last Measurement (AUC0-last) of MK-8583
Description: Values of plasma MK-8583 were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The area under the concentration time curve from time 0-last measurement (AUC0-last) of plasma MK-8583 is presented. The last quantified concentration value occurred at 2 hours (n=4) and 4 hours (n=1).
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr*nmol/L | 220 (415)

10. Secondary Outcome: Area Under the Concentration Time Curve From Time 0-infinity (AUC0-inf) of MK-8583
Description: Values of plasma MK-8583 were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: Due to insufficient plasma concentration data at the terminal phase, AUC0-inf of plasma MK-8583 was not able to be calculated for any participants. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Tmax of Plasma MK-8583.
Description: Values of plasma MK-8583 were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The time to achieve maximum concentration (Tmax) of plasma MK-8583 is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr. | 1 [0.5 to 2]

12. Secondary Outcome: Cmax of MK-8583
Description: Values of plasma MK-8583 were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The maximum concentration (Cmax) of plasma MK-8583 is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
nmol/L | 258 (440)

13. Secondary Outcome: t1/2 of MK-8583
Description: as for outcome 10
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: Due to insufficient plasma concentration data at the terminal phase, t1/2 of plasma MK-8583 was not able to be calculated for any participants. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 0

14. Secondary Outcome: Apparent Total Clearance (CL/F) of MK-8583
Description: Values of plasma MK-8583 were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The apparent total clearance (CL/F) of plasma MK-8583 is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: Due to insufficient plasma concentration data at the terminal phase, CL/F of plasma MK-8583 was not able to be calculated for any participants. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 0

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of MK-8583
Description: as for outcome 10
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: Due to insufficient plasma concentration data at the terminal phase, Vz/F of plasma MK-8583 was not able to be calculated for any participants. Participants from Panels B and C were not analyzed because they were not enrolled in the study.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 0

16. Secondary Outcome: AUC0-last of Tenofovir (TFV)
Description: Values of plasma TFV were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The area under the concentration time curve from time 0-last measurement (AUC0-last) of plasma TFV is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr*nmol/L | 1090 (187)

17. Secondary Outcome: AUC0-inf of TFV
Description: Values of plasma TFV were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The area under the concentration time curve from time 0-infinity (AUC0-inf) of plasma TFV is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr*nmol/L | 1550 (108)

18. Secondary Outcome: Tmax of TFV
Description: Values of plasma TFV were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The time to achieve maximum concentration (Tmax) of plasma TFV is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr. | 2 [1 to 4]

19. Secondary Outcome: Cmax of TFV
Description: Values of plasma TFV were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The maximum concentration (Cmax) of plasma TFV is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
nmol/L | 64.3 (137)

20. Secondary Outcome: t1/2 of TFV
Description: Values of plasma TFV were natural-log transformed and analyzed based on a linear model containing a fixed effect for the MK-8583 100-mg dose. The apparent terminal half-life (t1/2) of plasma TFV is presented.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.
Arm/Group | A: MK-8583 100mg
Number analyzed (Participants) | 5
hr. | 31.5 (13.2)

ADVERSE EVENTS:
Time Frame: Up to Day 29
Description: All participants who received at least one dose of treatment. Due to an earlier than anticipated achievement of the study objectives, a decision was made not to conduct Panels B and C.
Groups:
- MK-8583 100 mg: After fasting, a single oral dose of 100 mg MK-8583 in capsule form.
Arm/Group | MK-8583 100 mg | B: MK-8583 ≤ 150 mg | C: MK-8583 ≤ 150 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/5 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8583 100 mg (N=5) | B: MK-8583 ≤ 150 mg (N=0) | C: MK-8583 ≤ 150 mg (N=0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | NA | NA
Herpes zoster (Infections and infestations) | 1 (1) | NA | NA
Nasopharyngitis (Infections and infestations) | 1 (1) | NA | NA
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | NA | NA — Due to the nature of this Adverse Event and the small sample size for this study, the specific Adverse Event term for this Adverse Event is not disclosed due to patient confidentiality concerns.
Hepatic enzyme increased (Investigations) | 1 (1) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA
Haematoma (Vascular disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT03552536/Prot_SAP_000.pdf